CLINICAL TRIAL: NCT06434051
Title: The Effect of Traditional Chinese Cervical Manipulation for Cervicogenic Headache: a Pilot Randomized, Single-blind, Placebo-controlled Trial
Brief Title: Traditional Chinese Cervical Manipulation for Cervicogenic Headache
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, CHOW Chi Ho, Associate Professor of Practice, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Manipulation CGH
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Cervicogenic Headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Intervention Model Description: This intervention involves cervical mobilization that constitutes elements of cervical rotation and traction.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional Chinese cervical manipulation (Experimental): The CMP will first palpate the transverse processes of C1 and C2. The transverse process with apparent tenderness will be regarded as the pain side. The right side will be the painful side for the following example). During the manipulation, the CMP will use his left hand to support the lower jaw and passively rotate the neck to the left side by 70-75 degrees (or to the maximum angle without discomfort). The physician's right-hand fingers will support the left-side transverse processes of C1 and C2, and the thumb and thenar muscle will be placed on the spinous process and occipital area. While maintaining a passive left neck rotation, the physician will increase the rotation angle by 5-10 degrees with both hands under a sudden pulling force. The above procedure will be repeated on the right side (pain side).
  Interventions: Other: Traditional Chinese cervical manipulation
- Sham manipulation (Sham Comparator): The posture and position of the participant and the practitioner and the procedure are the same as the CCM technique. The right side will be regarded as the pain side once again. When performing the sham technique, the CMP uses the left hand to support the lower jaw position and passively rotates the neck to the left side by 70-75 degrees or to the maximum angle. The right hand presses the upper inner corner of the right scapula. While maintaining the passive left rotation of the neck, the right hand slowly exerts force downwards and outwards on the inner side of the scapula. The left hand only maintains the left rotation of the neck without any pulling force. After completion, repeat the above actions on the right side. After the technique is completed, participants can get up after resting for 5-10 minutes.
  Interventions: Other: Sham manipulation

INTERVENTIONS:
Other: Traditional Chinese cervical manipulation — The CMP will first palpate the transverse processes of C1 and C2. The transverse process with apparent tenderness will be regarded as the pain side. The right side will be the painful side for the following example). During the manipulation, the CMP will use his left hand to support the lower jaw and passively rotate the neck to the left side by 70-75 degrees (or to the maximum angle without discomfort). The physician's right-hand fingers will support the left-side transverse processes of C1 and C2, and the thumb and thenar muscle will be placed on the spinous process and occipital area. While maintaining a passive left neck rotation, the physician will increase the rotation angle by 5-10 degrees with both hands under a sudden pulling force. The above procedure will be repeated on the right side (pain side).
  Arms: Traditional Chinese cervical manipulation
Other: Sham manipulation — The posture and position of the participant and the practitioner and the procedure are the same as the CCM technique. The right side will be regarded as the pain side once again. When performing the sham technique, the CMP uses the left hand to support the lower jaw position and passively rotates the neck to the left side by 70-75 degrees or to the maximum angle. The right hand presses the upper inner corner of the right scapula. While maintaining the passive left rotation of the neck, the right hand slowly exerts force downwards and outwards on the inner side of the scapula. The left hand only maintains the left rotation of the neck without any pulling force. After completion, repeat the above actions on the right side. After the technique is completed, participants can get up after resting for 5-10 minutes.
  Arms: Sham manipulation

SUMMARY:
Background Cervical spondylosis is a prevalent condition. Studies has shown that it is a leading cause for headache, which is termed cervicogenic headache (CGH). The prevlance of CGH among severe headache is 17.5%. While conventional treatments, such as physical therapy and surgery, is effective in controlling symptoms, the effect was found to be short-lasting. There is existing clinical evidence supporting traditional Chinese cervical manipulation (CCM) as a viable treatment for CGH.

Objective To preliminarily assess the feasibility, safety, and effectiveness of CCM on patients with CGH, and to optimize parameters for a future large-scale trial.

Method This study is a pilot randomized, controlled, single-blind trial. 84 participants will be randomized evenly to receive either CCM or sham manipulation for 4 weeks. Outcome measurements will be conducted at baseline, week 2, week 4 and week 8 on cervical functional disability, cervical range of motion, and data on headache onset and painkiller assumption. Adverse events will be recorded using the Common Terminology Criteria for Adverse Events (CTCAE).

ELIGIBILITY:
Inclusion Criteria:

1. The diagnostic criteria of cervical spondylosis according to "The expert consensus on the classification, diagnosis, and non-surgical treatment of cervical spondylosis (2018)" are as follows:

   1. Patients must have a chief complaint of abnormal sensations such as pain in the occipital, neck, or shoulder area, and can be accompanied by related localized pain and tenderness
   2. X-ray imaging shows degenerative changes in the cervical spine
   3. Other conditions that could cause symptoms of the neck are excluded
2. The diagnostic criteria of CGH as listed by ICHD-3:

   a. Any headache fulfilling criterion C b. Clinical and/or imaging evidence of a disorder or lesion within the cervical spine or soft tissues of the neck, known to be able to cause headache c. Evidence of causation demonstrated by at least two of the following: i. headache has developed in temporal relation to the onset of the cervical disorder or appearance of the lesion ii. headache has significantly improved or resolved in parallel with improvement in or resolution of the cervical disorder or lesion iii. cervical range of motion is reduced and headache is made significantly worse by provocative manoeuvre iv. headache is abolished following diagnostic blockade of a cervical structure or its nerve supply v. Not better accounted for by another ICHD-3 diagnosis
3. Of age between 18 to 65 years old
4. Headache recurs for at least three months
5. The frequency of headaches in the past three months is at least once a week
6. The frequency, dosage, and type of painkillers have remained stable over the past 6 weeks
7. Score at least 10 points on the Neck Disability Index -

Exclusion Criteria:

1. Presented with red flag presentations of headache listed in the SNNOOP10 list (systemic symptoms/signs and disease, neurologic symptoms or signs, onset sudden or onset after the age of 40 years, and change of headache pattern), including fever, vascular and non-vascular intracranial diseases, history of brain tumor, brain neurological dysfunction or disorder, etc.
2. With suspected cervical spinal stenosis, cervical spinal cord lesions, cervical vascular disease, cervical nerve root disease, cervical instability, or cervical fracture
3. Has suffered from a whiplash injury within the past 6 weeks
4. Had surgery on the neck or head
5. Currently pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) scoring | Baseline, week 2, week 4 and week 8
  It is used to evaluate cervical functional disability It has good reliability and validity, reflecting the degree of limitation on living ability and the impact on quality of life. The higher the score, the more severe the symptoms.

SECONDARY OUTCOMES:
Active cervical range of motion | Baseline, week 2, week 4 and week 8
  to evaluate the range neck flexion, extension, left and right lateral flexion, left and right rotation. The measuring instrument will be the cervical goniometer.
Online headache diary: | Baseline, week 2, week 4 and week 8
  All participants are required to complete an online headache diary daily. It will include the following items: the time of headache onset, duration, pain intensity, and the type and frequency of painkillers taken

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Hong Kong Baptist University, Hong Kong
  - Lui Seng Chun,119 Lai Chi Kok Road, Mong Kok, Hong Kong

IPD SHARING:
Plan to Share IPD: No